CLINICAL TRIAL: NCT03823534
Title: Post-Op Pain Control for Prophylactic Intramedullary Nailing.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, David D. Greenberg, MD; Professor, Professor, Orthopaedic Surgery, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 28927
Record Dates: First submitted 2019-01-22; First posted 2019-01-30 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Bone Metastases; Lymphoma; Multiple Myeloma; Opioid Use; Pain
Keywords: Toradol; Ketorolac; Prophylactic intramedullary nail; bone metastases; Opioid use; post-operative pain
MeSH Terms: conditions — Lymphoma; Multiple Myeloma; Pain; Pain, Postoperative | interventions — Ketorolac; Ketorolac Tromethamine; Saline Solution; Acetaminophen; oxycodone-acetaminophen; Morphine; Oxycodone

STUDY DESIGN:
Intervention Model Description: This study is a prospective, randomized, double-blind, placebo-controlled trial.
Who Masked: Participant, Investigator
Masking Description: Both the patient and study investigators will be blinded. The hospital pharmacy will be unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Arm (Experimental): For the first 24 hours following surgery, patients younger than 65 years old will be administered a maximum of 120 mg/day bolus IV ketorolac (30 mg every 6 hours). Patients older than 65 years old or with history of advanced renal impairment will receive a maximum of 60 mg/day bolus IV ketorolac (15 mg every 6 hours). All patients may also be given acetaminophen 500 mg PO Q4 hours PRN for mild pain, oxycodone-acetaminophen 5-325 mg PO Q4 hours PRN for moderate- severe pain, and morphine IV PRN (or other opioid) for severe breakthrough pain while hospitalized. At discharge, they will be prescribed 1-2 hydrocodone-acetaminophen 5-325 mg Q4 hours, quantity 50. Those with preexisting liver disease will be prescribed the equivalent in oxycodone and will not receive acetaminophen for mild pain.
  Interventions: Drug: Ketorolac; Drug: Acetaminophen; Drug: Oxycodone Acetaminophen; Drug: Morphine; Drug: Hydrocodone/Acetaminophen; Drug: Oxycodone
- Control (Placebo Comparator): Following surgery, patients will be given acetaminophen 500 mg PO Q4 hours PRN for mild pain, oxycodone-acetaminophen 5-325 mg PO Q4 hours PRN for moderate-severe pain, and morphine IV PRN (or other opioid) for severe breakthrough pain while hospitalized. They will also be given a placebo injection of normal saline every 6 hours for the first 24 hours following surgery. At discharge, patients will be prescribed 1-2 hydrocodone-acetaminophen 5-325 mg Q4 hours PRN quantity 50, unless they have preexisting liver disease, in which case they will be prescribed the equivalent in oxycodone. They will not receive a nerve block.
  Interventions: Drug: Normal saline; Drug: Acetaminophen; Drug: Oxycodone Acetaminophen; Drug: Morphine; Drug: Hydrocodone/Acetaminophen; Drug: Oxycodone

INTERVENTIONS:
Drug: Ketorolac — IV Ketorolac to be given over the course of the first 24 hours after surgery. See arm/group description for further details.
  Other Names: Toradol
  Arms: Experimental Arm
Drug: Normal saline — An IV normal saline placebo prepared by the hospital pharmacy.
  Other Names: Placebo
  Arms: Control
Drug: Acetaminophen — acetaminophen 500 mg PO Q4 hours PRN for mild pain
  Other Names: Tylenol
Drug: Oxycodone Acetaminophen — oxycodone-acetaminophen 5-325 mg PO Q4 hours PRN for moderate to severe pain
  Other Names: Percocet
Drug: Morphine — morphine IV PRN (or other opioid) for severe breakthrough pain
Drug: Hydrocodone/Acetaminophen — At discharge, patients will be prescribed 1-2 hydrocodone-acetaminophen 5-325 mg Q4 hours. Those with preexisting liver disease will be prescribed the equivalent in oxycodone.
  Other Names: Norco
Drug: Oxycodone — Upon discharge, patients will be prescribed the equivalent of 1-2 hydrocodone 5mg Q4 hours upon should they have preexisting liver disease and are unable to consume acetaminophen.

SUMMARY:
Nationally, the opioid crisis has become a major epidemic with increasing mortality rates each year. Orthopedic surgeons routinely prescribe narcotics instead of NSAIDs for post-op pain control because of risk of delayed healing and nonunion due to NSAID use. Orthopedic oncology, however, has a unique subset of patients that undergo prophylactic placement of intramedullary femoral nails. Because no fracture is present, these patients do not rely on inflammatory healing factors, allowing for post-op NSAID use. This study sets out to determine the effect of post-op toradol use in addition to opioids compared to solely opioids in patients undergoing prophylactic nailing of the femur.

DETAILED DESCRIPTION:
Nationally, the opioid crisis has become a major epidemic with increasing mortality rates each year. Orthopedic surgeons routinely prescribe narcotics instead of NSAIDs for post-op pain control because of risk of delayed healing and nonunion due to NSAID use. Orthopedic oncology, however, has a unique subset of patients that undergo prophylactic placement of intramedullary femoral nails, often due to bone metastases that increase risk for future fractures. Because no fracture is present, these patients do not rely on inflammatory healing factors, allowing for post-op NSAID use.

Recent literature has demonstrated the efficacy of multi-modal pain management in treating post-op pain [1]. Currently, patients that undergo prophylactic intramedullary femur nail placement at SLU are often treated with both narcotics and toradol, as long as they can tolerate NSAIDs. However, the effect of toradol in addition to narcotics has not been determined. This study sets out to determine the effect of post-op toradol use in addition to opioids compared to solely opioids in patients undergoing prophylactic nailing of the femur.

ELIGIBILITY:
Inclusion Criteria:

1. Femoral Shaft or Neck bone lesion
2. 18 years old or greater
3. Plan to undergo prophylactic intramedullary nailing of one femur

Exclusion Criteria:

1. Concurrent pathologic fracture
2. History of advanced renal impairment (eGFR<30mL/min)
3. History of Peptic Ulcer Disease with bleeding or requiring hospitalization
4. History of NSAID or aspirin allergy
5. Concurrent chemotherapy regimen that prevents NSAID use
6. History of liver disease that precludes use of toradol
7. History of heart failure or cardiovascular disease that precludes toradol usage
8. Pregnancy
9. History of narcotic allergy resulting in anaphylaxis
10. Patients with coagulation disorders or those who require concomitant use of anticoagulant or anti- platelet therapy during the treatment phase of the study.
11. Patients with acetaminophen allergies resulting in anaphylaxis
12. Current use of the medication probenecid
13. Current use of the medication Pentoxifylline
14. History of aspirin induced asthma.
15. Known history of opioid dependence, abuse, or addiction.
16. Bilateral IMN of the femurs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-02-20 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Milligram Morphine Equivalent (MME) of Opioid Medications Utilized | Post-op days 1-14
  Measure the effect of post-op ketorolac on the concurrent use of opioid pain medications during post-op days 1-14 following prophylactic IMN of the femur compared to patients treated only with opioids.

SECONDARY OUTCOMES:
Patient Reported Outcomes Measurement System (PROMIS) Pain Intensity Scale | Up to six weeks post-op
  Measure the effect of post-op ketorolac on PROMIS Pain Intensity score compared to the PROMIS of those that receive only opioids. Total scores are computed by summing the scores of the 3 individual questions. Possible scores range from 3-15 with higher values representing increasing pain over the previous 7 days.
Single Assessment Numerical Evaluation (SANE) | Up to six weeks post-op
  Measure the effect of post-op ketorolac on SANE score compared to the SANE of those that receive only opioids. The score ranges from 0-100, with 100 representing the best possible perceived function of the limb and 0 the worst possible perceived function. There are no sub-scales.
Numerical Rating Scale (NRS) | Up to six weeks post-op
  Measure the effect of post-op ketorolac on NRS score compared to the NRS of those that receive only opioids. Scores range from 0-10 with higher scores signifying increasing pain. There are no sub-scales.

CONTACTS AND LOCATIONS:
Overall Officials: David Greenberg, MD, Principal Investigator — St. Louis University
Locations (1):
- Saint Louis University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cepeda MS, Carr DB, Miranda N, Diaz A, Silva C, Morales O. Comparison of morphine, ketorolac, and their combination for postoperative pain: results from a large, randomized, double-blind trial. Anesthesiology. 2005 Dec;103(6):1225-32. doi: 10.1097/00000542-200512000-00018. PMID 16306736